CLINICAL TRIAL: NCT06223620
Title: A Multicenter Retrospective Review of Management Strategies in Small Bowel Obstruction
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 046.GME.2018.D
Record Dates: First submitted 2023-10-18; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: SBO - Small Bowel Obstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: review performance of water soluble contrast — review performance of water soluble contrast study in patients admitted with SBO, will improve quality and safety, and decrease length of stay and morbidity.

SUMMARY:
The objective of the study is to review performance of water soluble contrast study in patients admitted with Small Bowel Obstruction(SBO), will improve quality and safety, and decrease length of stay and morbidity.

DETAILED DESCRIPTION:
Performance of contrast study has been a part of the protocols at multiple institutions of the southwestern surgical congress. Plan to perform a retrospective review of management protocols at these institutions. Wish to know whether the implementation of a standardized, protocol-driven pattern of practice involving the performance of water soluble contrast study in patients admitted with SBO, will improve quality and safety, and decrease length of stay and morbidity.

The objective of the study is to review performance of water soluble contrast study in patients admitted with SBO, will improve quality and safety, and decrease length of stay and morbidity.

Performance of contrast study has been a part of the protocols at multiple institutions of the southwestern surgical congress.

Hypothesize that implementation of a standardized, protocol-driven pattern of practice involving the performance of water soluble contrast study in patients admitted with SBO, will improve quality and safety, and decrease length of stay and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-89 years of age

  * Patients presenting with SBO

Exclusion Criteria:

* • Prisoners

  * Pregnant women

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previous studies found on an average 3.9 to 9.4% patient suffer from SBO. The disease incidence varies depending on the cause of obstruction. Assuming that 3.9% of the patients will be affected by SBO, the study would require a sample size of 504 for estimating the expected proportion with 3% absolute precision and 95% confidence.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Morbidity and length of stay | 1 year
  Morbidity and length of stay

SECONDARY OUTCOMES:
Patient demographics | 1 year
  number of patients (age, sex, weight, height)
admit date | 1 year
  Number of patients admitting to the hospital
discharge date | 1 year
  number of patients discharging
admission service | 1 year
  Number of services related to admissions
Aspirin(ASA )class | 1 year
  number of aspirin class
comorbidities | 1 year
  number of comorbidities associated
surgical history | 1 year
  number of surgeries in the past
labs | 1 year
  number of labs done
time of contrast given | 1 year
  rate of Contrast given

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No